CLINICAL TRIAL: NCT01496599
Title: Imaging Biomarkers in Parkinson Disease
Brief Title: Imaging Biomarkers in Parkinson s Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120031; 12-N-0031
Record Dates: First submitted 2011-12-17; First posted 2011-12-21 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01-27

CONDITIONS: Parkinson Disease
Keywords: Brain Imaging; Parkinson's Disease; Parkinsonism; Natural History; Parkinson Disease; PD; Healthy Volunteer; HV
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Volunteers: Subjects without PD diagnosis
- Parkinsons Disease subjects: Subjects fitting the MSD Clinical Diagnostic Criteria for PD
- Prodromal Parkinson disease: Subjects fitting the MDS prodromal criteria for PD

SUMMARY:
Background:

- Parkinson s disease (PD) causes slow movement, stiffness, and tremor. It results from the loss of a brain chemical called dopamine. PD gets worse over time, but researchers do not fully understand why the brain cells that produce dopamine stop working or die in people with PD. This study will use different ways of imaging the brain and brain chemicals to look at PD. It will compare brain imaging in people who definitely have PD to people who might have PD and to people without signs of PD. It will provide more information how the brain in people with PD changes over time.

Objectives:

- To understand the changes that occur in the brains of people with Parkinson s disease.

Eligibility:

* Individuals at least 18 years of age who have definite or possible Parkinson s disease.
* Healthy volunteers at least 18 years of age.

Design:

* Participants will have a screening visit with a physical exam and medical history.
* Participants will visit the National Institutes of Health Clinical Center every 18 month or 3 years for up to 9 years. There will be up to 6 total visits. Most visits will last 5 to 6 hours a day for 1 to 3 days.

Some or all of the following tests will be performed at each visit:

* Magnetic resonance imaging to take pictures of the brain. Some of these tests will be done at rest. Others will require participants to perform an activity during the scan.
* Medication withdrawal for 12 hours overnight for people taking PD medications. This may be done before some scans. Participants who feel unwell when they stop taking medications will be allowed to start taking them again.
* Participants will continue with the follow up visits until the end of the study.

DETAILED DESCRIPTION:
Objectives:

The purpose of this protocol is to evaluate possible imaging biomarkers for diagnosis and assessment of disease progression in Parkinson disease (PD) through multi-modal neuroimaging studies.

The study will have two parts:

1. Part 1: Compare brain images of PD subjects and healthy volunteers (HVs) using various imaging techniques in a case-control analysis.
2. Part 2: Compare findings on serial brain images with clinical assessments of clinically defined PD subjects, subjects with prodromal Parkinson disease, and healthy volunteers, over the following 9 years. The findings from this exploratory study will help develop additional hypothesis-driven studies investigating PD pathology. PD patients will yield information about how imaging outcomes change over time, and their relationship with disease progression; the patients with prodromal symptoms will give information as to which imaging modalities/analysis might predict the clinical manifestation of PD, healthy volunteers will serve as controls for subjects aging and technological changes due to scanner functioning.

   Study Population:

   Part 1 (Case-control study): 38 patients fitting the MSD Clinical Diagnostic Criteria for PD, and 38 age-matched healthy volunteers (HVs) as controls.

   Part 2 (Longitudinal study): We will continue to study qualifying subjects from Part 1 periodically over the following 9 years. We will also study 38 subjects fitting the MDS prodromal criteria for PD for up to 9 years.

   Design:

   Part 1: (Case-control study). Eligible participants will come for a 1 to 3 day visit. They will have a clinical assessment, and a magnetic resonance (MR) scans.

   Part 2: (Longitudinal study).

   -Participants will be followed up for up to 9 years. Each visit will last 2-3 days, during which they will have several outpatient tests done. Visits will be scheduled according to the following plan:

   --Subjects without neurological disorder (HV) will be seen every three years for a

   total of 9 years.

   --Subjects with clinical PD for more than 5 years will be seen every three years for a

   total of 9 years.
   * Subjects with clinical PD for less than 5 years will be seen every 18 months, until the 5y of diagnosis, and every three years after, for a total of 9 years.
   * Subjects assigned to the Prodromal group will be seen will every 18 months, until the 5y of diagnosis if symptoms do not progress into neurodegeneration (up to 3 visits), and until year 9 if symptoms progress towards PD.

     * Subjects who participated in the cross-sectional part will be included in the longitudinal section if they fulfill the inclusion/exclusion criteria. New subjects can be enrolled to complete this section.

   Outcome Measures:

   Primary outcome measures:
   * Structural MRI (SWI images): The primary outcome measure is the difference in susceptibility changes in iron-rich structures (ie. The SN, red nucleus, striatum) across groups and within groups over time.
   * Clinical presentation: We will evaluate how the prodromal symptoms influence the progression to clinical PD.

   Secondary outcome measures:
   * Structural MR (morphometry and diffusion analyses): The outcome measures are the differences in gray and white matter morphometry across groups and within groups over time. We will derive measures such as fractional anisotropy, trace, and parenchymal volume fractions as measures of fiber tract integrity, across groups and within groups over time.
   * fMRI: The outcome measure for fMRI is the difference in resting state functional connectivity patterns as reflected by BOLD signal fluctuations and their dynamics across groups and over time.
   * MRS: The outcome measure for MRS is the difference in the spectroscopy signal amplitude of phosphorus-containing compounds and neurotransmitters in the sensorimotor cortices and basal ganglia across groups and over time.

ELIGIBILITY:
* INCLUSION CRITERIA:

For all subjects:

* Age 18 or older.
* Subjects must fulfill either the clinically defined PD, prodromal PD or not having any of the red flags following the MDS criteria for PD.
* Able to give informed consent or, if there is evidence of cognitive decline, able to appoint a durable power of attorney (DPA) who can give informed consent.

EXCLUSION CRITERIA:

* More than 7 alcoholic drinks a week for females or 14 alcoholic drinks a week for males.
* History of a neurologic disorder such as a brain tumor, stroke, central nervous system infection, multiple sclerosis, a movement disorder other than the ones under study, epilepsy or a history of seizures or any abnormal or focal finding on neurological exam other than that associated with those studied in this protocol.
* History of any head injury with loss of consciousness
* Pregnancy or positive pregnancy test before the research procedure due to the risks associated with MRI scans. This would exclude subjects from participating in the protocol at that time.
* Inability to lie flat on the back for up to 2 hours
* Claustrophobia or a feeling of discomfort from being in small, enclosed spaces.
* Surgically or traumatically implanted metallic foreign bodies, such as pacemakers, implanted medical pumps, implanted hearing aids, metal plates in the skull or metal implants in the skull or eyes (other than dental fillings) that may be physically hazardous during an MRI, or might distort the images.
* Ablative surgery or implanted electrodes and generator for deep brain stimulation
* Use of the following therapies which may affect mitochondrial function: Coenzyme Q10, vitamin E, vitamin C, anti-retroviral drugs, chemotherapeutic agents, anti-epileptics agents or antibiotics. (Use ofthese substances will prevent getting MRS scan only).
* Have uncontrolled head movements that may impair image data collection

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Part 1 (Case-control study): We will study 30 patients with well-defined PD, as defined by the UK Parkinson s Society Brain Bank diagnostic criteria (Hughes et al., 1992, Olanow et al., 2009, Defer et al., 1999). We will also study 15 age-matched healthy volunteers (HVs) as controls. Part 2 (Longitudinal study): We will continue to study subjects from Part 1 periodically over the following 9 years. We will also study 30 subjects with early parkinsonism (EP). EP subjects are defined as individuals who have experienced at least one but fewer than 3 of the cardinal symptoms of PD at the time of enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2012-01-24 (Actual)

PRIMARY OUTCOMES:
Using MRI, we will measure signal intensities of iron-rich structures using T2 sequences and calculate phase shift values in these structures with susceptibility weighted sequences. We will also measure clinical symptom severity with the UPDRS s... | 10 years
  -Structural MRI (SWI images): The primary outcome measure is the difference in susceptibility changes in iron-rich structures (ie. The SN, red nucleus, striatum) across groups and within groups over time.-Clinical presentation: We will evaluate how the prodromal symptoms influence the progression to clinical PD.

SECONDARY OUTCOMES:
Structural MR (morphometry and diffusion analyses) | 10 years
  The outcome measures are the differences in gray and white matter morphometry across groups and within groups over time. We will derive measures such as fractional anisotropy, trace, and parenchymal volume fractions as measures of fiber tract integrity, across groups and within groups over time.
fMRI | 10 years
  The outcome measure for fMRI is the difference in resting state functional connectivity patterns as reflected by BOLD signal fluctuations and their dynamics across groups and over time.
MRS | 10 years
  The outcome measure for MRS is the difference in the spectroscopy signal amplitude of phosphorus-containing compounds and neurotransmitters in the sensorimotor cortices and basal ganglia across groups and over time.

CONTACTS AND LOCATIONS:
Overall Officials: Silvina G Horovitz, Ph.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share IPD and data dictionaries that underlie results in a publication. The data sharing will be restricted to those subjects whom have agreed to data sharing, and those authorized by the IRB if re-consenting were not an option.
Supporting Information: CSR
Time Frame: Starting 1 year after publication.
Access Criteria: IPD will be shared with qualified investigators, if allowed by IRB@@@@@@Any request for data sharing will be first reviewed by the protocol PI. @@@@@@The request must include the proposed use of the data. When requested data has IRB approval for data sharing, and the PI considers it a reasonable request, a memo of understanding will be signed by the parts, including the allowed use for the data. This will be done in consultation with the office of Tech Transfer.

REFERENCES:
- [Background] Narendra DP, Jin SM, Tanaka A, Suen DF, Gautier CA, Shen J, Cookson MR, Youle RJ. PINK1 is selectively stabilized on impaired mitochondria to activate Parkin. PLoS Biol. 2010 Jan 26;8(1):e1000298. doi: 10.1371/journal.pbio.1000298. PMID 20126261
- [Background] Olanow CW, Stern MB, Sethi K. The scientific and clinical basis for the treatment of Parkinson disease (2009). Neurology. 2009 May 26;72(21 Suppl 4):S1-136. doi: 10.1212/WNL.0b013e3181a1d44c. PMID 19470958
- [Background] Schapira AH. Mitochondria in the aetiology and pathogenesis of Parkinson's disease. Lancet Neurol. 2008 Jan;7(1):97-109. doi: 10.1016/S1474-4422(07)70327-7. PMID 18093566
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-N-0031.html